CLINICAL TRIAL: NCT07023289
Title: A Phase 2, Randomized, Open-Label Study Comparing Telisotuzumab Adizutecan (ABBV-400) Monotherapy to the Current Standard of Care in Subjects With Post Adjuvant ctDNA Positive Colorectal Cancer and No Radiographic Evidence of Disease (NED)
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity in Adult Participants Receiving Intravenously Infused Telisotuzumab Adizutecan Alone or With Standard of Care in Participants With Post Adjuvant Circulating Tumor DNA Positive Colorectal Cancer and No Radiographic Evidence of Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-534; 2024-518015-19-00 (Other: EU CT)
Record Dates: First submitted 2025-06-10; First posted 2025-06-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Telisotuzumab Adizutecan; ABBV-400, Stand of Care; Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Telisotuzumab Adizutecan Monotherapy (Experimental): Participants will receive telisotuzumab adizutecan dose A as a monotherapy, during the approximately 51 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Standard of Care (SOC) (Active Comparator): Participants will receive SOC, during the approximately 51 month study duration.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Arms: Telisotuzumab Adizutecan Monotherapy
Drug: Standard of Care — Standard of care treatment based on investigator's judgement to the active surveillance.
  Arms: Standard of Care (SOC)

SUMMARY:
Colorectal cancer (CRC) is the third most common type of cancer diagnosed worldwide. The purpose of this study is to assess change in disease activity when telisotuzumab adizutecan is given alone compared to standard of care (SOC) given alone.

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of CRC. This study will be divided into two groups called treatment arms. In arm 1 participants will receive telisotuzumab adizutecan alone. In arm 2 participants will receive SOC alone. Approximately 140 adult participants with CRC will be enrolled in the study in 45 sites worldwide.

In arm 1, participants will receive intravenous (IV) doses of telisotuzumab adizutecan alone. In arm 2 Participants will receive SOC alone. The study will run for a duration of approximately 51 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed adenocarcinoma of the colon or rectum.
* Surgical tumor material should be available and must be submitted for Signatera personalized panel and assessment of c-Met protein levels.
* Must have received at least 3 months of platinum-based doublet adjuvant chemotherapy but may not have been treated with topoisomerase inhibitors as part of adjuvant therapy.
* Has no radiographic evidence of disease (NED) confirmed by chest, abdominal, and pelvic computed tomography (CT) scans within 6 weeks prior to Cycle 1 Day 1 (C1D1) dosing.
* Circulating tumor deoxyribonucleic acid (ctDNA) positive after the end of adjuvant therapy and begin the treatment within 6 weeks after ctDNA is confirmed (reported).
* For participants with rectal cancer a total of at least 3 months of perioperative and/or adjuvant platinum-based doublet must have been administered. Please note that short course radiation or long-course chemoradiation does not count towards this 3-month minimum of platinum-doublet perioperative and/or adjuvant therapy.
* For participants with oligometastatic disease a total of at least 3 months of perioperative and/or adjuvant platinum-based doublet therapy must have been administered.

Exclusion Criteria:

* No availability of surgical tissue sample.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, or any evidence of active ILD or pneumonitis on screening chest computed tomography (CT) scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with disease free survival (DFS) Event | Up to Approximately 51 Months
  DFS is defined as the time from randomization to the time of first occurrence of first radiographic recurrence of colorectal cancer (CRC), (either local recurrence or distant metastases) as determined by the investigator, or death from any cause.

SECONDARY OUTCOMES:
Change in Circulating Tumor Deoxyribonucleic Acid (ctDNA) Clearance at 6 months | 6 Months
  ctDNA clearance at 6 months is defined as ctDNA negative at 6 months after randomization.
Overall Survival (OS) | Up to Approximately 51 Months
  OS is defined as the time from randomization to the event of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (16):
  - Providence Medical Foundation /ID# 274207, Fullerton, California
  - USC Norris Comprehensive Cancer Center /ID# 274550, Los Angeles, California
  - Mayo Clinic Hospital Jacksonville /ID# 274472, Jacksonville, Florida
  - University of Chicago Medical Center /ID# 274742, Chicago, Illinois
  - Johns Hopkins Hospital /ID# 275645, Baltimore, Maryland
  - University Of Michigan /ID# 273511, Ann Arbor, Michigan
  - Scri Minnesota Oncology Hematology, P.A. /ID# 275149, Minneapolis, Minnesota
  - Mayo Clinic-Rochester /ID# 273508, Rochester, Minnesota
  - Northwell Health Center for Advanced Medicine. /ID# 275331, Lake Success, New York
  - Northwest Cancer Specialists /ID# 275151, Portland, Oregon
  - SCRI Oncology Partners /ID# 274522, Nashville, Tennessee
  - Texas Oncology - Central/South Texas /ID# 275154, Austin, Texas
  - Texas Oncology-Grapevine /ID# 275155, Grapevine, Texas
  - The University of Texas MD Anderson Cancer Center /ID# 273539, Houston, Texas
  - Inova Schar Cancer Institute - Fairfax - Innovation Park Drive /ID# 274586, Fairfax, Virginia
  - Virginia Cancer Specialists - Fairfax /ID# 274339, Fairfax, Virginia
- Denmark (3):
  - Aarhus Universitetshospital - Skejby /ID# 274498, Aarhus, Central Jutland
  - Odense University Hospital /ID# 274970, Odense C, Region Syddanmark
  - Vejle Sygehus /ID# 274368, Vejle, Region Syddanmark
- Italy (3):
  - Azienda Ospedaliero Universitaria Careggi /ID# 273604, Florence, Firenze
  - IRCCS Istituto Clinico Humanitas /ID# 273566, Rozzano, Lombardy
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 273540, Naples, Napoli
- Japan (6):
  - Kyushu University Hospital /ID# 273710, Fukuoka, Fukuoka
  - Gifu University Hospital /ID# 274179, Gifu, Gifu
  - Yokohama City University Medical Center /ID# 273657, Yokohama, Kanagawa
  - Tohoku University Hospital /ID# 275481, Sendai, Miyagi
  - National Hospital Organization Osaka National Hospital /ID# 274306, Osaka, Osaka
  - Shizuoka Cancer Center /ID# 275480, Sunto-gun, Shizuoka
- South Korea (3):
  - Seoul National University Hospital /ID# 274451, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 274454, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 274452, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Hospital Universitario Virgen del Rocio /ID# 273720, Seville, Sevilla
  - Hospital Universitario La Paz /ID# 273718, Madrid
  - Hospital Universitario de Salamanca /ID# 273719, Salamanca
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 273745, Kaohsiung City
  - China Medical University Hospital /ID# 274644, Taichung
  - National Taiwan University Hospital /ID# 273580, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-534